CLINICAL TRIAL: NCT06552338
Title: The Wellness of Students Enrolled in Osteopathic Medical Schools Through Medical School and Residency Training
Brief Title: Wellness of Osteopathic Medical Students Throughout Their Training (Well-COM)
Acronym: Well-COM
Status: Recruiting | Type: Observational
Sponsor: Sam Houston State University (Other)
Responsible Party: Principal Investigator, Patrick Davis, Director of Research, Sam Houston State University
Other Study IDs: IRB-2024-217
Record Dates: First submitted 2024-07-25; First posted 2024-08-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Students, Medical
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Class of 2028
  Interventions: Other: Observational
- Class of 2029
  Interventions: Other: Observational
- Class of 2030
  Interventions: Other: Observational
- Class of 2031
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No intervention. Study is observational

SUMMARY:
The Well-COM Research Project addresses a critical gap in our understanding of the holistic health of medical students, over the entirety of the medical school experience. While the rigorous demands of medical education and its effects on the well-being of medical students are well-documented, there is a lack of long-term study assessing the mental, physical, and metabolic health of medical students from entry into medical school through their training and into residency. By collecting holistic health data from new first-year medical students, and over a minimum period of 10 years, the Well-COM project aims to provide invaluable insights into the changes in health and wellness experienced by medical students, thereby informing future interventions and support systems to promote overall health and resilience in medical school students.

ELIGIBILITY:
Inclusion Criteria:

* Medical student enrolled in SHSU college of osteopathic medicine.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Target population is students enrolled in osteopathic medical school
Sampling Method: Non-Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2025-12-07 (Estimated); Primary Completion 2034-12 (Estimated); Study Completion 2044-12 (Estimated)

PRIMARY OUTCOMES:
Burnout Index | Change over 10 years
  Maslach Burnout Inventory
Quality of Life Survey | Change over 10 years
  Short Form 8
Physical Fitness VO2 max | Change over 10 years
  Submaximal Step Test
Body Fat Percentage | Change over 10 years
  Portion of body mass composed of fat which is measure by bioelectrical impedance
Handgrip strength | Change over 10 years
  Maximal grip strength measured by a handgrip dynamometer
Total cholesterol | Change over 10 years
  Total cholesterol mg/dL
Blood pressure | Change over 10 years
  Systolic and diastolic blood pressure
Perceived Stress | Change over 10 years
  Perceived stress scale (PSS) Range 0-40 with higher scores indicating higher stress
Physical Activity | Change over 10 years
  The International Physical Activity Questionnaires (IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Davis, Principal Investigator — Sam Houston State University
Locations (1):
- Sam Houston State University College of Osteopathic Medicine, Conroe, Texas, United States

IPD SHARING:
Plan to Share IPD: No